CLINICAL TRIAL: NCT04717804
Title: 4D(Dimensional) CBCT (Cone-beam Computed Tomography) and Intrafractional Imaging for the Determination of the Most Representative 4D Simulation Planning Technique for Lung SBRT (Stereotactic Body Radiation Therapy) Technique Patients
Brief Title: 4D CBCT and Intrafractional Imaging for the Determination of the Most Representative 4D Simulation Planning Technique for Lung SBRT Technique Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CTMS# 20-0107
Record Dates: First submitted 2021-01-11; First posted 2021-01-22 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Cancer of Lung
MeSH Terms: conditions — Lung Neoplasms | interventions — Postmortem Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AIP (Average Intensity Projection) CT (Computed Tomagraphy) (Active Comparator): An image taken over a longer time of the lungs (average intensity projection of 4DCT) will be compared with breathing during treatment.
  Interventions: Other: AIP CT
- FB (Free-Breathing) CT (Placebo Comparator): A snapshot of breathing (free-breathing traditional CT) will be used to compare with breathing during treatment.
  Interventions: Other: FB (Free-Breathing) CT

INTERVENTIONS:
Other: AIP CT — An image taken over a longer time of the lungs (average intensity projection of 4DCT) will be compared with breathing during treatment.
  Other Names: CT Imaging
  Arms: AIP (Average Intensity Projection) CT (Computed Tomagraphy)
Other: FB (Free-Breathing) CT — A snapshot of breathing (free-breathing traditional CT) will be used to compare with breathing during treatment.
  Other Names: CT Imaging
  Arms: FB (Free-Breathing) CT

SUMMARY:
The researchers plan to investigate two ways of visualizing and planning to account for the respiratory motion which takes place while treating lung tumors with radiation therapy. The researchers will determine if a traditional snapshot (free-breathing) CT or a longer-lasting CT encompassing the breathing cycle better matches a patient's breathing during treatment.

DETAILED DESCRIPTION:
As part of this study the patient will receive the standard of care treatment of Stereotactic Body Radiation Therapy (SBRT) approach for treatment of lung cancer. The study will compare whether the quick snapshot or longer-last image is more representative of breathing motion. The standard of care way to verify breathing is to use the Cone Beam Computerized Tomography (CBCT) before each treatment. For this study the researchers will use two other standard of care ways to verify breathing motion during treatment only during the first and last radiation treatment sessions. During the other radiation treatment sessions the CBCT alone will be used. These two other methods are FDA approved, but not routinely being used at the Mays Cancer Center. One method is called 4D-CBCT and is conducted immediately prior to treatment. This will create an image taken over a longer time of the patient's lungs which will be compared with the images from the CT Simulation used to plan the radiation. The other way is called Intrafractional CBCT and is imaging that is done at the same time as the radiation treatment delivery. This will show the researchers how the tumor is moving while the radiation treatment is taking place. These two methods require a longer treatment time, approximately 10 minutes during the first and last treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Ability to provide informed written consent in either English or Spanish.
* Patients with cancer or presumed cancer involving the lung (primary or secondary) planned to undergo lung SBRT technique or IMRT technique with an SBRT setup in 10 or fewer fractions.

Exclusion Criteria:

* Current pregnancy, as this is a contraindication to receiving radiation therapy.
* Patients to be treated to multiple targets concurrently.
* Any condition or history as evidenced by patient record and/or self-report that, in the opinion of the investigator, would interfere with adherence to the prescribed pattern of radiation therapy.
* Poor lung function, as judged by the prescribing radiation oncologist, sufficiently limiting to make the patient not a candidate for 4D imaging (for example major differences between the 4D and free-breathing CT scan).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
To investigate radiation therapy treatment tumor localization accuracy by determining whether the FB or AIP images is more representative of the target at treatment. | 2 weeks
  This will be quantitively determined by quantifying the agreement between the two CT scans using the Dice coefficient (DSC) as a metric for localization accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Saenz, PhD, Principal Investigator — UT Health San Antonio
Locations (1):
- Mays Cancer Center, UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No